CLINICAL TRIAL: NCT02791802
Title: A European Multicenter Study on the Effect of Lipoprotein(a) Elimination by Lipoprotein Apheresis on Cardiovascular Outcomes
Brief Title: Effect of Lipoprotein(a) Elimination by Lipoprotein Apheresis on Cardiovascular Outcomes
Acronym: MultiSELECt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Collaborators: Kaneka Pharma Europe N.V. (Industry)
Responsible Party: Principal Investigator, Prof. Bernd Hohenstein, Prof. Dr. med. Bernd Hohenstein, Technische Universität Dresden
Other Study IDs: TUD-LPA16-001
Record Dates: First submitted 2016-05-26; First posted 2016-06-07 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Lipoprotein Types--Lp System Lp(A) Hyperlipoproteinemia
Keywords: Lipoprotein(a); lipoprotein/lipid apheresis; CV disease
MeSH Terms: conditions — Lipoprotein Types--Lp System Lp(A) Hyperlipoproteinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For biosampling one additional serum (9 ml), one EDTA vaccutainer (2.7 ml) and two PAXgene™ Blood RNA Tubes and 10 ml Urine samples will be provided for each subject.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A: Lipoprotein apheresis subjects: Established cardiovascular disease with disease progression indicated by one major cardiovascular event. With or without subsequent cardiovascular events/interventions, despite adequately controlled cardiovascular risk factors occuring within the last 2 years prior to enrolment. Corrected Low-density lipoprotein cholesterol < 100 mg/dL (2.6 mmol/l) during 3 months prior to study enrolment.
  Additional lipoprotein apheresis is established following enrolment using the following established systems: Dextran-sulfate adsorption (DSA) from plasma and whole blood, Heparin-induced LDL precipitation apheresis (HELP®), Polyacrylate adsorption from whole blood and simple DFPP (DALI® and Monet®), ApoB100-immunoadsorption (TheraSorbLDL®, Temperature-optimized double filtration plasmapheresis (DFPP).
- Group B: Control group: Established cardiovascular disease with disease progression indicated by one major cardiovascular event. With or without subsequent cardiovascular events/interventions, despite adequately controlled cardiovascular risk factors occuring within the last 2 years prior to enrolment. Corrected Low-density lipoprotein cholesterol < 100 mg/dL (2.6 mmol/l) during 3 months prior to study enrolment.
  The control group will not undergo a sham apheresis procedure. It is an open trial.

SUMMARY:
This multicenter multinational prospective two-arm matched-pair observational study aims to establish a prospective comparison of active lipoprotein apheresis treatment approved and conducted according to German guidelines for the indication of elevated Lp(a) versus a maximum tolerated lipid-lowering therapy as standard care. Due to the prospective character and the inclusion of a control arm, this will be the first clinical study that can confirm the relevance of the established approach to use lipoprotein apheresis in those subjects and its effects to reduce the individual cardiovascular risk. The optimized management of subjects in the control group (not receiving lipoprotein apheresis) will also help to clarify the controversial issue, to which extent intensive medical care per se can influence the occurence of subsequent cardiovascular events. Primary objective of the trial is to evaluate the clinical benefit of Lp(a) reduction using lipoprotein apheresis on myocardial infarction, PCI, CABG, fatal and non- fatal stroke, transient ischemic attack, interventional or surgical revascularization of peripheral arteries and death from cardiovascular disease. The primary objective of this study evaluates the clinical benefit of weekly lipoprotein apheresis in subjects with progressive cardiovascular disease, as accepted by the German Federal Joint Committee as indication for subjects with elevated Lp(a). Comparator will be matched subjects under maximum tolerated lipid lowering therapy without access to lipoprotein apheresis treatment. The clinical benefit will be defined as the reduction of the composite endpoint of major adverse cardiovascular events (MACE), defined as either myocardial infarction, PCI, CABG, fatal and non-fatal stroke, transient ischemic attack or death from cardiovascular disease over a period of at least 2 years after completion of visit 1b and until at least 60 events of the primary end-point occurred in group B. If the number of at least 60 documented primary endpoint events within 2 years of the completion of enrolment did not occur, the study will continue until this number of primary endpoint events has accumulated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 70
2. Male or female
3. Written informed consent
4. Lipoprotein(a) > 60 mg/dL, or > 120 nmol/L using an alternative laboratory method
5. Corrected Low-density lipoprotein cholesterol < 100 mg/dL (2.6 mmol/l) during 3 months prior to study enrolment.
6. Established cardiovascular disease with disease progression indicated by one major cardiovascular event, which might be either

   * myocardial infarction
   * PCI
   * CABG
   * Stroke
   * or revascularization of peripheral arteries using PTA, stenting or bypass surgery

   (with or without subsequent cardiovascular events/interventions) despite adequately controlled cardiovascular risk factors* occuring within the last 2 years prior to enrolment

   (*Hypertension, Diabetes, tobacco consumption, LDL Cholesterol)
7. Platelet aggregation inhibitors or systemic anticoagulation according to cardiologic indication
8. Positive recommendation by central Trial Expert Committee

Exclusion Criteria:

1. Previous lipoprotein apheresis therapy
2. Triglyceride concentrations ≥ 250 mg/dL (2.8 mmol/L)
3. Known homozygous or compound heterozygous familial hypercholesterolemia
4. Known type III hyperlipoproteinemia
5. Pregnancy, breast feeding
6. Active smoking, defined as any inhaled tobacco consumption with in the last 3 months
7. Uncontrolled hypertension (>160/90 mmHg)
8. Active malignant disease
9. Planned major surgical procedures
10. Current participation in an interventional trial
11. Contraindication for apheresis therapy (e. g. necessity of ACE inhibitor therapy)
12. CKD stages IV and V
13. Diabetes mellitus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants have to be 18 years or older and need to be intellectually capable to understand and follow the study protocol. All subjects have to present with progressive cardiovascular disease and need to fulfill the criteria fixed in the recommendations by the German Joint Federal Committee (in German: "Gemeinsamer Bundesausschuss"; see section 1.2). In addition, a TEC has to verify presence of the treatment indication and will be blinded with respect to subject's group assignment. Apheresis subjects (group A) will be included in chronological order, since this will most likely reflect the natural distribution of disease in the general population. Control subjects (group B) will then be matched to the lipoprotein apheresis subjects entering the study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-08; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The primary end-point is an at least 10 % reduction of the proportion of events | 2 years of follow-up
  The primary end-point is an at least 10 % reduction of the proportion of events regarding the composite end-point consisting either of myocardial infarction, PCI, CABG, fatal and non-fatal stroke, transient ischemic attack, interventional or surgical revascularization of peripheral arteries or death from cardiovascular disease (or any combination of these) at the final visit.

SECONDARY OUTCOMES:
An at least 10 % reduction of the proportion of events | 2 years of follow-up
  An at least 10 % reduction of the proportion of events regarding the composite endpoint of cardiovascular death, major coronary event, cerebrovascular accidents and stroke.
An at least 10 % reduction of the proportion of events | 2 years of follow-up
  An at least 10 % reduction of the proportion of events regarding the composite endpoint of cardiovascular death, major coronary events and all cerebrovascular events.
An at least 10 % reduction of the proportion of events regarding the composite Secondary endpoints of the Trial | 2 years of follow-up
  An at least 10 % reduction of the proportion of events regarding the composite endpoint of CV death, non-fatal MI, documented unstable angina that requires admission into a hospital, all revascularization (including both coronary and non-coronary) occurring at least 30 days after the MACE event, the rate of in-stent restenosis and non-fatal stroke.

OTHER OUTCOMES:
Reduction of individual endpoints | 2 years of follow-up
  Reduction of individual endpoints at the final visit, reported as % reduction of the number of cumulated and individual events
  * death from any cause,
  * CHD death,
  * CV death,
  * MI,
  * documented unstable angina that requires admission into a hospi-tal,
  * all coronary revascularization occurring at least 30 days after a prior MACE event:
    * either PCI or
    * CABG
  * all revascularization (including both coronary and non-coronary) occurring at least 30 days after a prior MACE event,
  * in-stent restenosis rate,
  * stroke,
  * transient ischemic attack,
  * Percentage of subjects achieving a mean reduction of Lp(a) of 60% or more
  * Mean reduction of Lp(a)
  * Percentage of subjects achieving mean LDL-C reduction of 60 % or more
  * Number of apheresis related side effects
  * Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Hohenstein, MD, Principal Investigator — Technische Universität Dresden
Locations (12):
- Germany (12):
  - University Hospital Carl Gustav Carus, Dresden, Saxony
  - Herz- und Diabeteszentrum NRW Universitätsklinik der Ruhr-Universität Bochum Klinik für Kardiologie, Bad Oeynhausen
  - Dialyse am Kortumpark, Bochum
  - Nephrologisches Zentrum Göttingen, Göttingen
  - PHV Dialysezentrum, Meißen
  - Klinikum der Universität München Campus Innenstadt, München
  - Klinikum der Universität München Campus Großhadern, München
  - Dialysezentrum Potsdam, Potsdam
  - Nierenzentrum Reinbek, Reinbek
  - Nephrocare Rostock GmbH Medizinisches Versorgungszentrum Südstadt, Rostock
  - Nephrologisches Zentrum, Villingen-Schwenningen
  - Heinrich Braun Klinikum, Zwickau

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study Homepage — http://www.multiselect-trial.eu